CLINICAL TRIAL: NCT05863091
Title: Respiratory Rate Validation Study With Accuracy Analysis of Respiratory and Breathing Pattern Extracted by Impedance Change of Patch-type Electrocardiogram Device (HiCardi+ Wearable Patch Device, Mezoo Co., Ltd.)
Brief Title: Respiratory Rate Validation Study - HiCardi+ Wearable Patch Device, Mezoo Co., Ltd.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1-2022-0055
Record Dates: First submitted 2023-04-19; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis; Asthma
Keywords: Pulmonary Function Testing(PFT); Ventilator; Patch-type electrocardiogram device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group of patients undergoing pulmonary function tests (Experimental): Patients undergoing pulmonary function tests with spontaneous breathing
  Interventions: Device: HiCardi+
- A group of patients on ventilators in an intensive care unit (Experimental): Among patients who are on a ventilator, those on the Richmond agitation sedation scale -4 to -5 and who do not breathe spontaneously
  Interventions: Device: HiCardi+

INTERVENTIONS:
Device: HiCardi+ — A patch-type electrocardiogram device is attached to a patient undergoing pulmonary function tests.
  Arms: A group of patients undergoing pulmonary function tests
Device: HiCardi+ — A patch-type electrocardiogram device is attached to a patient on a ventilator in an intensive care unit.
  Arms: A group of patients on ventilators in an intensive care unit

SUMMARY:
The purpose of this study is to analyze the accuracy of respiratory and breathing patterns generated through impedance changes generated by a patch-type electrocardiogram device (HiCardi+ wearable patch device, Mezoo Co., Ltd.), targeting patients undergoing pulmonary function testing and ventilator application.

DETAILED DESCRIPTION:
Subjects The target number of participants for this study is 211, consisting of 181 patients undergoing pulmonary function testing and 30 patients using a ventilator.

* Spontaneous breathing subjects (181 patients): Assuming that a pulmonary function testing examiner with spontaneous breathing would examine about 50 patients per day, a total of 181 subjects will be targeted, taking into consideration the possibility of refusals.
* Non-Spontaneous breathing subjects (30 patients): In addition, in the case of patients with a Richmond Agitation Sedation Scale of -4 to -5 who use a ventilator and do not have spontaneous breathing, the final 30 subjects will be conducted for the purpose of data collection for about 6 hours.

Focus of the study The tidal volume and respiratory amplitude will be analyzed in detail through pulmonary function tests, and the respiratory rate will be analyzed through ventilator data.

Study method The study method is as follows: In the pulmonary function testing room, consent will be obtained from patients undergoing pulmonary function testing, and a patch-type electrocardiogram device will be attached before the test is conducted. The records of the ECG patch generated during the approximately 30-minute pulmonary function test and the results of the pulmonary function test will be acquired. Based on the impedance obtained from the patch-type electrocardiogram, the pulmonary function test results are extracted as the reference data related to the respiratory pattern. Correlation analysis is performed on the tidal volume and respiratory amplitude obtained through this comparison. Additionally, Bland-Altman analysis is conducted on the validation set, which is divided into an 8:2 training set and validation set, for the algorithm that predicts tidal volume and respiratory amplitude.

For patients with RASS -4 to -5 who are on a ventilator, the patch-type electrocardiogram device is attached for about 6 hours after the consent of the patient caregiver, and the data generated from the ECG patch and the ventilator are compared and analyzed. Based on the impedance obtained from the patch-type electrocardiogram, the data from the ventilator will be used as reference data related to respiratory rate. Mean Difference (MD), Standard Deviation (SD), degrees of freedom (df), bias, regression, and limits of agreement will be calculated through correlation analysis and Bland-Altman analysis on the obtained respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 and older

Exclusion Criteria:

* patients under the age of 19
* patients cannot apply the patch-type electrocardiogram device due to physical defects or contact allergic reactions
* patients do not consent to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate measured by pulmonary function test | During the pulmonary function test (about 30 minutes)
  The respiratory rate will be analyzed for correlation and Bland-Altman analysis using continuous variables generated from pulmonary function testing, ventilator information, and patch-type ECG device. Mean difference (MD), standard deviation (SD), degrees of freedom (df), bias, regression, and limits of agreement will be calculated.
Respiratory rate measured by ventilator | about 6 hours
  The respiratory rate will be analyzed for correlation and Bland-Altman analysis using continuous variables generated from pulmonary function testing, ventilator information, and patch-type ECG device. Mean difference (MD), standard deviation (SD), degrees of freedom (df), bias, regression, and limits of agreement will be calculated.
Respiratory rate measured by patch-type electrocardiogram device | up to 6 hours
  The respiratory rate will be analyzed for correlation and Bland-Altman analysis using continuous variables generated from pulmonary function testing, ventilator information, and patch-type ECG device. Mean difference (MD), standard deviation (SD), degrees of freedom (df), bias, regression, and limits of agreement will be calculated.

SECONDARY OUTCOMES:
Tidal volume measured by pulmonary function test, ventilator, and patch-type electrocardiogram device | -Pulmonary function test: During the pulmonary function test (about 30 minutes) -Ventilator application: about 6 hours
  For tidal volume and respiratory amplitude, correlation analysis is performed on continuous variables generated from pulmonary function tests, ventilator information, and a patch-type electrocardiogram measuring device. Additionally, the algorithm for predicting respiratory volume and respiratory amplitude is divided into a training set and a validation set in an 8:2 ratio, and Bland-Altman analysis is performed on the validation set.
respiratory amplitude measured by pulmonary function test, ventilator, and patch-type electrocardiogram device | -Pulmonary function test: During the pulmonary function test (takes about 30 minutes) -Ventilator application: about 6 hours
  For tidal volume and respiratory amplitude, correlation analysis is performed on continuous variables generated from pulmonary function tests, ventilator information, and a patch-type electrocardiogram measuring device. Additionally, the algorithm for predicting respiratory volume and respiratory amplitude is divided into a training set and a validation set in an 8:2 ratio, and Bland-Altman analysis is performed on the validation set.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea